CLINICAL TRIAL: NCT05146297
Title: Diversity and Inclusion in Research Underpinning Trials
Brief Title: Diversity and Inclusion in Research Underpinning Prevention and Therapy Trials
Acronym: DISRUPT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Nina Bickell, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 21-0012
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Liver Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Liver Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Participants (Active Comparator): Patients with invasive breast, prostate or liver cancer, who face a treatment decision
  Interventions: Behavioral: Clinical trial match-list
- Physician Participants (Active Comparator): Oncologists, and advanced practitioners caring for patients with breast, prostate, liver cancer including medical, surgical, radiation oncologists, interventional radiologists, urologists & hepatologists
  Interventions: Behavioral: Match-list intervention

INTERVENTIONS:
Behavioral: Clinical trial match-list — Creation and dissemination educational materials designed to inform and empower patients' participation in their cancer treatment including the consideration of clinical trial participation and provide clinical trials' patient navigators (CTPN) to further aid with education about clinical trials.
  Arms: Patient Participants
Behavioral: Match-list intervention — Providers by intervening at the clinical and systems levels to provide them with tools and processes and informational and practical support to facilitate CT consideration, discussion, and offer to aid with education about clinical trials and facilitate CT consideration at a treatment decision node.
  Arms: Physician Participants

SUMMARY:
This proposal brings together multidisciplinary teams from four New York City institutions charged with reducing cancer disparities that affect approximately two million people residing in some of the most diverse and underserved communities in the United States. The intent of this collaborative research is captured by its acronym, DISRUPT: Diversity & IncluSion in Research Underpinning Prevention & Therapy Trials. To disrupt the norms that maintain heightened risk and poorer outcomes experienced by BIPOC, the research team propose three integrated and synergistic aims to improve diversity and inclusion in CTs through disruptive approaches at the community (Aim 1), provider, system and patient (Aim 2), and basic and translational scientist levels (Aim 3). All three aims focus on metrics for changing norms reified in institutional policies and established practice that will provide essential evidence to translate and scale these changes to institutions and networks involved in cancer treatment research. In Aim 1, the research team will partner with local organizations to formulate and disseminate new norms regarding cancer care and research and diffuse these new norms throughout the community via community organizations and Health Ambassadors bringing a different vantage point on CTs, raising awareness and increasing demand for access to cancer research. In Aim 2, the research team will create an electronic approach to identify key clinical characteristics of patients and trials and match patients and trials and bring these data to patients and their physicians at the time of key decisions. In Aim 3, the research team will provide and integrate essential experiential training in diversity, social determinants of health and the importance of conducting community-relevant work into basic and translational science training. This DISRUPT proposal provides the foundation to disrupt norms about cancer clinical trials in our communities, delivery systems and scientific research enterprises.

ELIGIBILITY:
Inclusion Criteria:

* All patients >21 years of age with invasive breast, lung or liver cancer, who face a treatment decision
* patients of doctors who have consented to participate
* able to give consent and speak either English or Spanish
* For provider recruitment, oncologists, and advanced practitioners caring for patients with breast, lung, liver cancer including medical and surgical oncologists, interventional radiologists & hepatologists will be eligible

Exclusion Criteria:

* Patients who are unable to give consent
* unable to understand English or Spanish
* lack of invasive breast/liver cancer
* those who do not face an imminent treatment decision

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Trial Accrual | from start to the conclusion of recruitment to the clinical trial, average of 2 months
  Change in rates of clinical trial accrual of the total population and BIPOC population.

SECONDARY OUTCOMES:
Number of physicians agree to usefulness of the match lists | at 6 months post intervention implementation
  Number of physicians who find the match lists useful to inform decision-making and clinical trial participation.
Patient Post-intervention Survey | 2 weeks post intervention implementation
  Survey is not summed: there is no scoring or a scale for survey. Questions will be looked at individually for statements related to patient level barriers that influenced CT discussions and offers. Some answers are yes/no while others may multiple choices.
Physician Post -intervention survey | at 6 months post intervention implementation
  Survey is not summed: there is no scoring or a scale for survey. Questions will be looked at individually for statements related to patient, physician, and system level barriers that influenced CT discussions and offers. Some answers are yes/no while others may multiple choices.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bickell, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Herbert Irving Comprehensive Cancer Care Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
undecided

REFERENCES:
- [Derived] Bickell NA, May B, Havrylchuk I, John J, Lin S, Tao A, Yagnik R, Tatonetti NP. Implementation of a rule-based algorithm to find patients eligible for cancer clinical trials. JAMIA Open. 2024 Nov 18;7(4):ooae131. doi: 10.1093/jamiaopen/ooae131. eCollection 2024 Dec. PMID 39559491